CLINICAL TRIAL: NCT06343233
Title: Multicenter, Prospective Observational Study of Patients Aged 65 Years or Older, Hospitalized for Acute Heart Failure.
Brief Title: FAiling HearT in the Elderly (FATE) Study
Acronym: FATE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Multimedica (Other)
Responsible Party: Sponsor
Other Study IDs: FATE
Record Dates: First submitted 2024-03-17; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Frailty
Keywords: heart failure; Fraility; ELderly; primary and secondary prevention
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: usual care — The aim is to set up a collection of clinical and instrumental data of usual care from patients hospitalized for acute heart failure aged ≥ 65; at the time of admission and after 6-12 and 18 months from the event (admission).

SUMMARY:
In 2015 the Italian Ministry of Health invited the Cardiac Research Hospitals of Italy to constitute a Cardiac Network. The aim of the network is to facilitate and promote scientific and technological research in the setting of cardiovascular diseases and related risk factors. The Cardiology Network, responding to the indications of the National Health Research Program, which includes research models oriented towards prevention studies with objectives and priority areas of intervention such as "acquiring scientific knowledge necessary for implementing both secondary and tertiary prevention programs for patients and primary prevention for contacts, where indicated, or for subjects exposed to specific risk factors", aims to identify strategies and/or prognostic and predictive factors of outcomes through the construction of thoroughly studied case series and systematic collection of biological materials, as well as the definition of research models based on clinical outcomes.

The Study aims to examine the impact of clinical practice and therapies, analytically considering treatments and other important covariates that contribute in a complex manner to the therapeutic success of patients with heart failure.

DETAILED DESCRIPTION:
Heart failure is a clinical condition continuously growing, characterized by an unfavorable prognosis both in terms of life and health. It is increasingly common and often associated with other clinical conditions that complicate its course, worsen the prognosis, and increase costs for the National Health Service (NHS). Heart failure (HF) is characterized by high prevalence (3% of the adult population, approximately 600,000 patients already diagnosed in Italy) and incidence (0.1-0.2, 87,000 cases/year). Patients with chronic HF may experience disease exacerbations leading to frequent hospitalizations, which, however, are appropriate in only a minority of cases.

Heart failure is a leading cause of death and hospitalization, especially in patients over 65 years of age. The annual incidence of heart failure doubles for every decade over 65 years, with a prevalence reaching 10% in patients over 80 years of age. Age is also one of the major determinants of prognosis in heart failure patients and is associated with a higher presence of comorbidities that contribute to worse outcomes. However, fewer data are available for patients over 65 years of age, who are often excluded from major clinical and pharmacological trials.The FATE Study considers the population presenting the most common disease pattern among hospitalized patients, particularly those with acute heart failure (AHF) and older age (> 65 years), in which the syndrome manifests with greater aggressiveness and complexity, also due to various frequently associated medical conditions. The study aims to provide clinical information in a broad sample that includes the subpopulation of patients who are usually not adequately represented in traditional clinical studies or even excluded, namely the elderly subjects. Therefore, the development of the FATE study will provide a unique tool for healthcare management methodologies. The study design will use highly flexible data collection strategies, particularly useful in the dynamics of data collection in patients.

The FATE Study considers the population presenting the most frequent disease pattern among hospitalized patients, particularly those with acute heart failure (AHF) and older age (> 65 years), in which the syndrome manifests with greater aggressiveness and complexity, also due to various frequently associated medical conditions. The study aims to provide clinical information in a broad sample that includes the subpopulation of patients who are usually not adequately represented in traditional clinical studies or even excluded, namely the elderly subjects. Therefore, the development of the FATE study will provide a unique tool for healthcare management methodologies. The study design will use highly flexible data collection strategies, particularly useful in the dynamics of data collection in patients. With its specific characteristics, the Study aims to examine the impact of clinical practice and therapies, analytically considering treatments and other important covariates that contribute in a complex manner to the therapeutic success of patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 65 years;
* Patients hospitalized for acute heart failure;
* Signature of informed consent.

Exclusion Criteria:

* Patients with significant valvular pathology at T0/Baseline (index event);
* Patients with malignant neoplasms or systemic pathology with a prognosis "quoad vitam" less than 1 year;
* Patients with known active infectious diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years or older hospitalized for acute decompensated heart failure (ADHF). The index event must be documented, at the time of discharge, by the need for intravenous administration of specific treatments and classified based on the International Classification of Diseases (ICD-9 code 428 or codes consistent with the presence of any heart failure, for primary or secondary disease).
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization or death at 12 months | up to 12 months
  Analyzing the prevalence of hospitalizations and/or deaths due to cardiovascular causes at 12 months from enrollment.

SECONDARY OUTCOMES:
Hospitalization or death at 6-12-18 months | up to 6-12-18 months
  Prevalence of hospitalizations and/or death from all causes at 6, 12, and 18 months from enrollment;
hospitalizations and/or death from cardiovascular causes | up to 6 and18 months
  Prevalence and incidence of hospitalizations and/or death from cardiovascular causes at 6 and 18 months;
association between events and patient characteristics | up to 18 months
  Analysis of the association between events (hospitalization and/or death) and clinical characteristics, instrumental findings, and patient co-pathologies. Both cardiovascular events and those occurring for all causes will be evaluated, stratifying the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gaia CAttadori, MD, Principal Investigator — MultiMedica - IRCCS MultiMedica - Cardiology
Locations (7):
- Italy (7):
  - Istituti clinici scientifici Maugeri - IRCCS Montescano ( Cardiologia DPT), Montescano, Italy/Pavia
  - IRCCS Centro Cardiologico Monzino, Milan, MIlano
  - IRCCS Humanitas Research Hospital, Rozzano, Milano
  - IRCCS MultiMedica, Sesto San Giovanni, Milano
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan
  - IRCCS Auxologico, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343
- [Result] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Result] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822
- [Result] Ezekowitz JA, O'Meara E, McDonald MA, Abrams H, Chan M, Ducharme A, Giannetti N, Grzeslo A, Hamilton PG, Heckman GA, Howlett JG, Koshman SL, Lepage S, McKelvie RS, Moe GW, Rajda M, Swiggum E, Virani SA, Zieroth S, Al-Hesayen A, Cohen-Solal A, D'Astous M, De S, Estrella-Holder E, Fremes S, Green L, Haddad H, Harkness K, Hernandez AF, Kouz S, LeBlanc MH, Masoudi FA, Ross HJ, Roussin A, Sussex B. 2017 Comprehensive Update of the Canadian Cardiovascular Society Guidelines for the Management of Heart Failure. Can J Cardiol. 2017 Nov;33(11):1342-1433. doi: 10.1016/j.cjca.2017.08.022. Epub 2017 Sep 6. PMID 29111106
- [Result] Krum H, Jelinek MV, Stewart S, Sindone A, Atherton JJ; National Heart Foundation of Australia; Cardiac Society of Australia and New Zealand. 2011 update to National Heart Foundation of Australia and Cardiac Society of Australia and New Zealand Guidelines for the prevention, detection and management of chronic heart failure in Australia, 2006. Med J Aust. 2011 Apr 18;194(8):405-9. doi: 10.5694/j.1326-5377.2011.tb03031.x. PMID 21495941